CLINICAL TRIAL: NCT04640415
Title: Continuous Wireless Monitoring of Vital Signs and Automated Alerts of Patient Deterioration vs. Routine Monitoring of High-risk Patients After Major Surgery. A Randomized Controlled Trial.
Brief Title: Continuous Wireless Monitoring of Vital Signs and Automated Alerts of Postsurgical Patient Deterioration.
Acronym: WARD-RCT-SX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Bispebjerg Hospital (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Jesper Mølgaard, MD, Ph.d student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-20034555
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Complication,Postoperative
Keywords: Wireless Monitoring; Vital signs; Physiologic deterioration
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No alarms (No Intervention): Patients will be connected to monitoring equipment, registering vital sign data, but data will be blinded to clinical staff.
- Active alarms (Active Comparator): Patients will be connected to monitoring equipment, registering data, and data will be available to clinical staff, including alarms for vital sign deterioration.
  Interventions: Device: Active Alarms

INTERVENTIONS:
Device: Active Alarms — Intervention consists of actively alerting staff personnel if physiologic vital signs, deviates from certain thresholds for more than a set duration. Continuous vital sign data will also be available to clinical staff.
  Arms: Active alarms

SUMMARY:
The primary aim of the current study is to assess the effect of continuous wireless vital sign monitoring with generation of real-time alerts, compared to blinded monitoring without alerts on the cumulative duration of any severely deviating vital signs in patients admitted to general hospital wards after major surgery.

We hypothesize that continuous vital signs monitoring, and real-time alerts will reduce the cumulative duration of severely deviating vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute or elective major abdominal (laparotomy/laparoscopy), major orthopedic, major urologic, or arterial vascular surgery.
* Estimated duration of surgery ≥2 hours and at least two expected overnight stays.
* Randomization and commencement of continuous wireless monitoring possible within 24 hours postoperatively

Exclusion Criteria:

* Patient expected not to cooperate with study procedures.
* Allergy to plaster or silicone.
* Impaired cognitive function (in uncertain cases assessed by a Mini Mental State Examination] score < 24)
* Patients admitted for palliative care only (i.e. no active treatment).
* Planned admission to unit using continuous vital sign monitoring (i.e. an intermediary care/telemetry unit).
* Patients previously enrolled in the medical WARD RCT.
* Patients with a pacemaker or Implantable Cardioverter Defibrillator (ICD) device.
* Inability to give informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Cumulative duration | During monitoring, for a maximum of up to 5 postoperative days or until discharge.
  Cumulative duration of one or more deviations in vital signs. List of vital signs, and normal limits detailed in protocol.

SECONDARY OUTCOMES:
Frequency of sustained deviation alerts | During monitoring, for a maximum of up to 5 postoperative days or until discharge.
  Frequency of each of the sustained deviations in vital signs. List of vital signs, and normal limits detailed in the protocol.
Any adverse event | 7 days and 30 days after start of monitoring
  Any adverse event. Criteria for each defined in protocol. Results will be compared between the case and control arm, on when it a diagnosis is made.
  Based on information in patient electronic medical file.
Any serious adverse event | 7 days and 30 days after start of monitoring
  Any serious adverse event. Criteria for each defined in protocol. Serious Adverse Events will be determined using the criteria as defined in ICH-GCP terms.
  Results will be compared between the case and control arm, on when it a diagnosis is made.
  Based on information in patient electronic medical file.

OTHER OUTCOMES:
Length of hospital stay | 30 postoperative days and 6 months
  Length of hospital stay
Patient related post-admission healthcare expenses | 2 years
  Total patient-related healthcare expenses in patients experiencing adverse clinical outcomes compared to patients without such outcomes and the effect of the study intervention on expenses
Staff response time (intervention group only) | During monitoring, for a maximum of up to 5 postoperative days or until discharge, whichever comes first
  Time from the staff is notified by app, until they respond by selecting 'check on patient' in app Stratified according to time of day

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Mølgaard, MD, Principal Investigator — Rigshospitalet, Denmark; Eske K Aasvang, MD, DMSc, Study Chair — Rigshospitalet, Denmark; Christian S Meyhoff, MD, PhD, Study Chair — Bispebjerg
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen NV, Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molgaard J, Gronbaek KK, Rasmussen SS, Eiberg JP, Jorgensen LN, Achiam MP, Rohrsted M, Singh UM, Hoang TH, Sogaard M, Meyhoff CS, Aasvang EK. Continuous Vital Sign Monitoring at the Surgical Ward for Improved Outcomes After Major Noncardiac Surgery: A Randomized Clinical Trial. Anesth Analg. 2025 Oct 1;141(4):807-817. doi: 10.1213/ANE.0000000000007606. Epub 2025 Jul 1. PMID 40591492
- See also: Related Info — http://www.ward247.com

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04640415/SAP_000.pdf